CLINICAL TRIAL: NCT00834977
Title: Randomized, 2-way, Crossover, Bioequivalence Study of Amlodipine-Benazepril 10mg-20mg Capsules and Lotrel® Administered as 1 x 10 Mg-20 mg Capsule in Healthy Subjects Under Fasting Conditions.
Brief Title: Amlodipine-Benazepril 10mg-20mg Capsules in Healthy Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 40012
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — benazepril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amlodipine Benazepril (Experimental): Amlodipine Benazepril 10mg-20mg Capsule (test) dosed in first period followed by Lotrel® 10mg-20mg Capsule (reference) dosed in second period
  Interventions: Drug: Amlodipine-benazepril 10 mg-20 mg capsules
- Lotrel® (Active Comparator): Lotrel® 10mg-20mg Capsule (reference) dosed in first period followed by Amlodipine Benazepril 10mg-20mg Capsules (test) dosed in second period
  Interventions: Drug: Lotrel® 10 mg-20 mg capsule

INTERVENTIONS:
Drug: Amlodipine-benazepril 10 mg-20 mg capsules — 1 x 10-20 mg
  Arms: Amlodipine Benazepril
Drug: Lotrel® 10 mg-20 mg capsule — 1 x 10-20 mg
  Arms: Lotrel®

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of amlodipine-benzazepril 10 mg-20 mg capsules (test) versus Lotrel® (reference), administered as 1 x 10 mg capsule under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Male of non-child-bearing potential female, non-smoker, 18 years of age and older.
* Non-child-bearing potential female subjects is defined as follows:
* Post-menopausal state: absence of menses for 12 months prior to drug administration or hysterectomy woth bilateral oophorectomy at least 6 months prior to drug administration.
* Surgically sterile: hysterectomy, bilateral oophorectomy, or tubal ligation at least 6 months prior to drug administration.
* Capable of consent

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks prior to the administration of the study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the Medical Sub-Investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judges clinically significant.
* Positive testing for hepatitis B, hepatitis C, or HIV at screening.
* EGC abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 100 ot over 140 nnHg, diastolic blood pressure lower than 60 or over 90 mmHg, or heart rate less that 60 or over 100 bpm) at screening.
* BMI ≥ 30.0
* History of significant alcohol abuse within six months prior to the screening visit or any indication of the regular use of more than fourteen units of alcohol per week ( 1 Unit= 150 mL of wine, 360 mL of beer, or 45 mL ot 40% alcohol) or positive alcohol breath test at screening.
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs( such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to the screening visit or positive urine drug screen at screening.
* History of allergic reactions to heparin,amlodipine,benazepril, or other ACE inhibitors, or other related drugs.
* Use of any drugs known to induce hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; examples of inhibitors: antidepressant (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to administration of the study medication.
* Use of and investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver of kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Any clinically significant history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric, or metabolic disease.
* Use of prescription medication ( including hormone replacement therapy) within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Difficulty to swallow study medication. Subjects who have used tobacco in any form within the 90 days preceding study drug administration
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the Medical Sub-Investigator, could contraindicate the subject's participation in this study.
* A depot injection or an implant of any drug within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 30 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows:
* 50 mL to 300 mL of whole blood within 30 days,
* 301 mL to 500 mL of whole blood within 45 days, or
* more than 500 mL of whole blood within 56 days prior to drug administration.
* Consumption of food or beverages containing grapefruit ( e.g. fresh, canned, or frozen) within 7 days prior to administration of the study medication.
* Intolerance to venipunctures
* Unable to understand or unwilling to sign the Informed Consent Form.
* Clinically significant history of angioedema. Subjects with a clinically significant history or active hypotension. Subjects with a significant history of active neutropenia and/or agranulocytosis.
* Breast-feeding subject.
* Positive urine pregnancy test at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-04; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, M.D., Principal Investigator — Anapharm
Locations (2):
- Canada (2):
  - Anapharm Inc., Montreal, Quebec
  - SFBC Anapharm, Sainte-Foy, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Amlodipine Benazepril (Test) First: Amlodipine Benazepril 10/20 mg capsule (test) dosed in first period followed by Lotrel® 10/20 mg capsule (reference) in second period
- Lotrel® (Reference) First: Lotrel® 10/20 mg capsule (reference) dosed in first period followed by Amlodipine Benazepril 10/20 mg capsule (test) dosed in second period
Period: First Intervention
Arm/Group | Amlodipine Benazepril (Test) First | Lotrel® (Reference) First
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Amlodipine Benazepril (Test) First | Lotrel® (Reference) First
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amlodipine Benazepril (Test) First | Lotrel® (Reference) First | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 21 | 44
  >=65 years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 16 | 17 | 33
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 1 | 1
  White | 21 | 20 | 41
  Hispanic | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  Canada | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Amlodipine
Description: Bioequivalence based on Cmax - Maximum observed concentration
Time Frame: Blood samples collected over 168 hour period
Population: One subject was excluded from all statistical analysis for Amlodipine based on a pre-dose plasma concentration greater than 5% of the Cmax value.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Amlodipine Benazepril: Amlodipine Benazepril 10/20 mg capsule (test) dosed in either period
- Lotrel®: Lotrel® 10/20 mg capsule (reference) dosed in either period
Arm/Group | Amlodipine Benazepril | Lotrel®
Number analyzed (Participants) | 47 | 47
pg/mL | 6299.49 (1917.69) | 6185.06 (1697.24)
Statistical Analysis 1: Comparison: Amlodipine Benazepril vs Lotrel®; Test type: Non-Inferiority or Equivalence — Parametric analysis of variance (ANOVA)on AUC0-t, AUCinf and Cmax; geometric Confidence Intervals for AUC0-t, AUC0-inf and Cmax; Ratio of Least Squares Means = 101.08, 90% CI [97.23 to 105.09] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

2. Primary Outcome: AUC0-inf - Amlodipine
Description: Bioequivalence based on AUC0-inf - Area under the concentration-time curve from time zero to infinity (extrapolated)
Time Frame: Blood samples collected over 168 hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Amlodipine Benazepril | Lotrel®
Number analyzed (Participants) | 47 | 47
pg*h/mL | 365612.90 (143713.73) | 366523.24 (140268.40)
Statistical Analysis 1: Comparison: Amlodipine Benazepril vs Lotrel®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 99.38, 90% CI [96.63 to 102.22] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

3. Primary Outcome: AUC0-t - Amlodipine
Description: Bioequivalence based on AUC0-t - Area under the concentration-time curve from time zero to time of last non-zero concentration (per participant)
Time Frame: Blood samples collected over 168 hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Amlodipine Benazepril | Lotrel®
Number analyzed (Participants) | 47 | 47
pg*h/mL | 328249.86 (118686.43) | 331782.17 (114025.75)
Statistical Analysis 1: Comparison: Amlodipine Benazepril vs Lotrel®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 98.48, 90% CI [95.80 to 101.23] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

4. Primary Outcome: Cmax - Benazepril
Description: Bioequvialence based on Cmax - Maximum observed concentration
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Amlodipine Benazepril | Lotrel®
Number analyzed (Participants) | 48 | 48
ng/mL | 330.93 (162.44) | 340.57 (163.48)
Statistical Analysis 1: Comparison: Amlodipine Benazepril vs Lotrel®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 98.72, 90% CI [86.95 to 112.09] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

5. Secondary Outcome: Cmax - Benazeprilat
Description: Cmax - Maximum observed concentration
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Amlodipine Benazepril | Lotrel®
Number analyzed (Participants) | 48 | 48
ng/mL | 378.27 (117.87) | 397.50 (126.07)
Statistical Analysis 1: Comparison: Amlodipine Benazepril vs Lotrel®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 95.69, 90% CI [90.54 to 101.14] — Metabolite presented for informational purposes only

6. Secondary Outcome: AUC0-inf - Benazeprilat
Description: AUC0-inf - Area under the concentration-time curve from time zero to infinity (extrapolated)
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Amlodipine Benazepril | Lotrel®
Number analyzed (Participants) | 48 | 48
ng*h/mL | 2027.53 (559.69) | 2033.12 (508.26)
Statistical Analysis 1: Comparison: Amlodipine Benazepril vs Lotrel®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Slope = 99.43, 90% CI [96.48 to 102.46] — Metabolite presented for informational purposes only

7. Primary Outcome: AUC0-inf - Benazepril
Description: Bioequivalence based on AUC0-inf - Area under the concentration-time curve from time zero to infinity (extrapolated)
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Amlodipine Benazepril | Lotrel®
Number analyzed (Participants) | 48 | 48
ng*h/mL | 245.15 (113.78) | 253.21 (125.50)
Statistical Analysis 1: Comparison: Amlodipine Benazepril vs Lotrel®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 97.20, 90% CI [92.82 to 101.78] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

8. Primary Outcome: AUC0-t - Benazepril
Description: as for outcome 3
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Amlodipine Benazepril | Lotrel®
Number analyzed (Participants) | 48 | 48
ng*h/mL | 241.65 (113.50) | 250.13 (125.21)
Statistical Analysis 1: Comparison: Amlodipine Benazepril vs Lotrel®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 96.99, 90% CI [92.52 to 101.68] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

9. Secondary Outcome: AUC0-t - Benazaprilat
Description: AUC0-t - Area under the concentration-time curve from time zero to time of last non-zero concentration (per participant)
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Amlodipine Benazepril | Lotrel®
Number analyzed (Participants) | 48 | 48
ng*h/mL | 1981.29 (556.26) | 1990.26 (506.70)
Statistical Analysis 1: Comparison: Amlodipine Benazepril vs Lotrel®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 99.24, 90% CI [96.21 to 102.35] — Metabolite presented for informational purposes only

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is not permitted to discuss or publish trial results.